CLINICAL TRIAL: NCT03092921
Title: The Evaluation of a Mask for the Treatment of Obstructive Sleep Apnea (OSA)
Brief Title: The Evaluation of a Mask Seal/Mask for the Treatment of Obstructive Sleep Apnea (OSA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIA-209
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Sleep Disordered Breathing; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- F&P Mask Seal (Experimental): Participants to use trial seal in-home for 1 week
  Interventions: Device: F&P Mask Seal
- F&P Mask (Experimental): Participants to use trial mask in-home for 2 weeks
  Interventions: Device: F&P Mask

INTERVENTIONS:
Device: F&P Mask Seal — Investigative Mask Seal to be used for OSA therapy
  Arms: F&P Mask Seal
Device: F&P Mask — Investigative Mask to be used for OSA therapy
  Arms: F&P Mask

SUMMARY:
This investigation is designed to evaluate the performance as well as the patients overall acceptance of the seal/mask.

DETAILED DESCRIPTION:
A minimum of 15 OSA participants who currently use a Full face mask will be recruited for the trial. Participant will be on the trial for 1 week- The participant will use the trial seal in-home for 1 week.

An additional 5 Participants will be added to the study to use the entire mask in home for 14+-4 days as an extension to the original trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18+ years of age)
* Able to give consent
* Apnea hypopnea Index (AHI)≥ 5 on diagnostic night
* Prescribed PAP for OSA
* Existing oro-nasal mask user

Exclusion Criteria:

* Inability to give consent
* Patients who are in a coma or a decreased level of consciousness
* Anatomical or physiological conditions making automatic positive airway pressure (APAP) therapy inappropriate (e.g. unconsolidated facial structure)
* Commercial drivers who are investigated by New Zealand Transport Agency
* Current diagnosis of carbon dioxide (CO2) retention
* Pregnant or may think they are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2017-08-03 (Actual); Study Completion 2017-08-03 (Actual)

PRIMARY OUTCOMES:
Ease of use | 1 week in home
  Subjective questionnaire
Acceptability | 1 week in home
  Subjective questionnaire
Ease of use | 2 weeks in home
  Subjective questionnaire
Acceptability | 2 weeks in home
  Subjective questionnaire

SECONDARY OUTCOMES:
Objective leak data | 1 week in home
  Obtained from participants' device

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Gunson, Principal Investigator — Employee
Locations (1):
- Fisher & Paykel Healthcare, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No
For product development purposes only. Data will be deidentified.